CLINICAL TRIAL: NCT00542789
Title: A Phase III, Multicentre, Randomised, Double-blind, Parallel-group, Comparative Efficacy and Safety Study of Esomeprazole(20 mg Once Daily) Versus Placebo for the Prevention of Gastric and/or Duodenal Ulcers Associated With Daily Nonsteroidal Anti-inflammatory Drug (NSAID) Use
Brief Title: Comparative Efficacy & Safety Study of Esomeprazole Versus Placebo for the Prevention of Gastric and Duodenal Ulcers With NSAID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D961HC00001
Record Dates: First submitted 2007-10-11; First posted 2007-10-12 (Estimated); Results first posted 2010-05-28 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2010-05

CONDITIONS: Gastric Ulcer; Duodenal Ulcer; Rheumatoid Arthritis; Osteoarthritis; Lumbago
Keywords: gastrointestinal; GI; NSAID; Japan; Japanese; Gastric ulcer; duodenal ulcer
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer; Arthritis, Rheumatoid; Osteoarthritis; Low Back Pain | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Experimental): Esomeprazole 20 mg
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole — 20mg once daily oral
  Other Names: Nexium
  Arms: 2
Drug: Placebo — once daily oral
  Arms: 1

SUMMARY:
The purpose of this study is to assess the efficacy of esomeprazole (D961H) 20 mg versus placebo once daily for up to 24 weeks of treatment involving patients with a history of gastric and/or duodenal ulcers receiving daily nonsteroidal anti-inflammatory drug (NSAID) therapy by evaluating presence or absence of gastric and/or duodenal ulcers throughout the treatment period (24 weeks) in terms of efficacy on prevention of gastric and/or duodenal ulcers

ELIGIBILITY:
Inclusion Criteria:

* Medical history of gastric and/or duodenal ulcer
* A diagnosis of a chronic condition (rheumatoid arthritis, osteoarthritis, lumbago,etc) that requires daily NSAID use,at least 20 years of age

Exclusion Criteria:

* Having gastric or duodenal ulcer in active or healing stage according to the Sakita/Miwa classification
* History of esophageal, gastric or duodenal surgery
* Having severe liver disease or chronic renal disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2007-08; Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naotsugu Oyama, Study Director — AstraZeneca Japan
Locations (39):
- Japan (39):
  - Research Site, Chiryū, Aichi-ken
  - Research Site, Seto, Aichi-ken
  - Research Site, Yotukaido, Chiba
  - Research Site, Miyaodai, Fukuoka
  - Research Site, Sapporo, Hokkaido
  - Research Site, Akashi, HYOGOi
  - Research Site, Itami, Hyōgo
  - Research Site, Koto, Hyōgo
  - Research Site, Nishinomiya, Hyōgo
  - Research Site, Hitachi, Ibaragi
  - Research Site, Morioka, Iwate
  - Research Site, Sagamihara, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kōtari, Kyoto
  - Research Site, Kyoto, Kyoto
  - Research Site, Chiisagata, Nagano
  - Research Site, Matsumoto, Nagano
  - Research Site, Nagano, Nagano
  - Research Site, Sasebo, Nagasaki
  - Research Site, Beppu, Oita Prefecture
  - Research Site, Ōita, Oita Prefecture
  - Research Site, Ibara, Okayama-ken
  - Research Site, Hirakata, Osaka
  - Research Site, Osaka, Osaka
  - Research Site, Sakai, Osaka
  - Research Site, Suita, Osaka
  - Research Site, Takatsuki, Osaka
  - Research Site, Kawagoe, Saitama
  - Research Site, Saitama, Saitama
  - Research Site, Fukuroi, Shizuoka
  - Research Site, Hamamatsu, Shizuoka
  - Research Site, Izunokuni, Shizuoka
  - Research Site, Maikinohara, Shizuoka
  - Research Site, Shizuoka, Shizuoka
  - Research Site, Yaizu, Shizuoka
  - Research Site, Shimotsuke, Tochigi
  - Research Site, Chiyoda City, Tokyo
  - Research Site, Koto, Tokyo
  - Research Site, Musashimurayama, Tokyo

REFERENCES:
- [Derived] Sugano K, Kinoshita Y, Miwa H, Takeuchi T; Esomeprazole NSAID Preventive Study Group. Randomised clinical trial: esomeprazole for the prevention of nonsteroidal anti-inflammatory drug-related peptic ulcers in Japanese patients. Aliment Pharmacol Ther. 2012 Jul;36(2):115-25. doi: 10.1111/j.1365-2036.2012.05133.x. Epub 2012 May 16. PMID 22591121

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 343 randomised participants 341 in Full Analysis set and safety analysis set. Full set used for summaries of baseline char. and efficacy variables. Safety set used for summaries of safety variables. 2 excluded, took no investigational drug or had protocol deviation. 173 Esomeprazole 20 and 168 placebo had baseline information and were summarised.
Pre-assignment Details: Out of 1246 enrolled participants, 343 participants were randomised and 903 participants were not randomised. The major reasons of no randomisation were 'Did not meet eligibility criteria' (877 participants) and 'Voluntary discontinuation by participant' (24 participants).
Groups:
- Experimental: Esomeprazole 20 mg: Esomeprazole 20 mg once daily oral
- Comparater: Placebo: Placebo once daily oral
Period: Overall Study
Arm/Group | Experimental: Esomeprazole 20 mg | Comparater: Placebo
Started | 175 (Randomised) | 168 (Randomised)
Completed | 134 | 90
Not Completed | 41 | 78
Not completed — Adverse Event | 18 | 17
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Protocol Violation | 8 | 1
Not completed — Recurrence of Gastric Ulcer | 8 | 57

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Esomeprazole 20 mg | Comparater: Placebo | Total
Number analyzed (Participants) | 175 | 168 | 343
Age, Customized [Number; unit: participants]
  <65 years | 78 | 91 | 169
  Between 65 and 74 years | 59 | 54 | 113
  >=75 years | 36 | 23 | 59
  Missing | 2 | 0 | 2
Sex/Gender, Customized [Number; unit: participants]
  Female | 108 | 100 | 208
  Male | 65 | 68 | 133
  Missing | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Absence of Gastric and/or Duodenal Ulcer Throughout the Treatment Period
Description: The absence of gastric and/or duodenal ulcer throughout the treatment period
Time Frame: each visit up to 24 weeks
Population: Two participants were excluded from these sets because they took no investigational drug or had major protocol deviation. As the result, the numbers of participants for gender baseline were 173 in Esomeprazole 20 mg and 168 in Placebo, respectively.
Measure: Number; unit: Participants
Arm/Group | Experimental: Esomeprazole 20 mg | Comparater: Placebo
Number analyzed (Participants) | 173 | 168
Participants | 167 | 112

2. Secondary Outcome: Absence of Gastric and/or Duodenal Ulcer up to 4 Weeks After Treatment
Description: The absence of gastric and/or duodenal ulcer up to 4 weeks after treatment
Time Frame: up to 4 weeks
Measure: Number; unit: Participants
Arm/Group | Experimental: Esomeprazole 20 mg | Comparater: Placebo
Number analyzed (Participants) | 173 | 168
Participants | 172 | 133

3. Secondary Outcome: Absence of Gastric and/or Duodenal Ulcer up to 12 Weeks After Treatment
Description: The absence of gastric and/or duodenal ulcer up to 12 weeks after treatment
Time Frame: up to 12 weeks
Measure: Number; unit: Participants
Arm/Group | Experimental: Esomeprazole 20 mg | Comparater: Placebo
Number analyzed (Participants) | 173 | 168
Participants | 168 | 119

ADVERSE EVENTS:
Arm/Group | Experimental: Esomeprazole 20 mg | Comparater: Placebo
Serious Adverse Events (participants affected / at risk) | 12/173 | 5/168
Other Adverse Events (participants affected / at risk) | 134/173 | 124/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Esomeprazole 20 mg (N=173) | Comparater: Placebo (N=168)
Colonic Polyp (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Faeces Discoloured (Gastrointestinal disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastroduodenal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Pneumonia Pneumococcal (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Pneumonia Bacterial (Infections and infestations) | 0 | 1
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small Intestine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Medical Device Complication (Injury, poisoning and procedural complications) | 1 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Esomeprazole 20 mg (N=173) | Comparater: Placebo (N=168)
Abdominal Pain Upper (Gastrointestinal disorders) | 18 | 22
Abdominal Distension (Gastrointestinal disorders) | 15 | 11
Stomach Discomfort (Gastrointestinal disorders) | 15 | 17
Nausea (Gastrointestinal disorders) | 11 | 9
Reflux Oesophagitis (Gastrointestinal disorders) | 10 | 13
Diarrhoea (Gastrointestinal disorders) | 9 | 6
Constipation (Gastrointestinal disorders) | 7 | 5
Dyspepsia (Gastrointestinal disorders) | 7 | 10
Nasopharyngitis (Infections and infestations) | 27 | 27
Pharyngitis (Infections and infestations) | 3 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 3
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 7 | 1
Anorexia (Metabolism and nutrition disorders) | 11 | 6
Hepatic Function Abnorma (Hepatobiliary disorders) | 6 | 1
Hypertension (Vascular disorders) | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other